CLINICAL TRIAL: NCT01222546
Title: Phase I, Open-label, Multi-center, Dose-escalation Study to Evaluate Safety, Pharmacokinetics and Activity of CH5132799 Administered Orally as a Monotherapy in Patients With Advanced Solid Tumors
Brief Title: Study of CH5132799 Administered Orally in Patients With Advanced Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Chugai Pharma Europe Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PA-001EU
Record Dates: First submitted 2010-10-14; First posted 2010-10-18 (Estimated); Last update posted 2014-06-23 (Estimated); Status verified 2014-06

CONDITIONS: Solid Tumors
MeSH Terms: interventions — CH 5132799

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- CH5132799 (Experimental)
  Interventions: Drug: CH5132799

INTERVENTIONS:
Drug: CH5132799

SUMMARY:
This is an open-label, multi-center, dose-escalation Phase I study to evaluate safety, pharmacokinetics and activity of CH5132799 administered orally as a single agent in patients with advanced solid tumors.

ELIGIBILITY:
Inclusion Criteria:

1. Provision of signed written informed consent.
2. Histologically or cytologically confirmed diagnosis of advanced solid tumor.
3. Age ≥ 18 years.
4. Eastern Cooperative Oncology Group (ECOG) performance status of 0, 1 or 2.
5. Life expectancy of ≥ 12 weeks.
6. Disease measurability:

   Patients must have a measurable - as per Response Evaluation Criteria in Solid Tumours (RECIST) criteria version 1.1 - and/or evaluable disease.
7. Paraffin-embedded archival tumor tissue available. Fresh biopsies will be required if no paraffin embedded tumor tissues available.
8. Adequate bone marrow function.
9. Adequate cardiac function: Patient should have Left Ventricular Ejection Fraction (LVEF) of ≥ 50% as determined by echocardiography (ECHO) or Multi Gated Acquisition (MUGA) scans.
10. Adequate liver function.
11. Adequate renal function.
12. Adequate adrenal function assessed by baseline cortisol of > 200 nmol/L
13. Ability to comply with protocol requirements.
14. Female patients must be postmenopausal (12 months of amenorrhea), surgically sterile or they must agree to use a physical method of contraception. Male patients who have been sterilized must agree to use a barrier method of contraception. Male subjects must also commit to use a barrier method of contraception until at least 3 months after the end of study treatment.
15. Female patients of child-bearing potential must have a negative serum pregnancy test within the seven days prior to the first study drug administration.

Exclusion Criteria:

1. History of allergic reactions attributed to components of the formulated product.
2. Inability to swallow oral medications or impaired gastrointestinal absorption due to active inflammatory bowel disease.
3. Known Central Nervous System (CNS) metastases or leptomeningeal metastases will be eligible only if it could be radiologically demonstrated that there is no CNS disease progression during the 3 months prior to the study
4. Known active or uncontrolled pulmonary dysfunction.
5. Uncontrolled hypertension
6. Prior chemotherapy, radiotherapy (other than short cycle of palliative radiotherapy for bone pain), or immunotherapy within 28 days of first receipt of study drug (within 6 weeks for nitrosoureas and mitomycin C). Hormone therapy within 14 days of first receipt of study drug, with exception of prostate cancer if indicated.
7. Prior toxicities from chemotherapy or radiotherapy which have not regressed to Grade ≤ 1 severity - National Cancer Institute Common Terminology Criteria for Adverse Events (NCI-CTCAE version 4.0).
8. Type 1 or 2 diabetes mellitus requiring regular medication and/or a fasting plasma glucose (FPG) ≥ 120 mg/dL (or 6.6 mmol/dL) at screening.
9. Increased QTc interval (QTc > 450 ms for male; > 460 ms for female).
10. History of heart failure, refractory hypokalemia to adequate supplementation, family history of long QT syndrome or other risk factors for "Torsades de Pointes", and/or the use of concomitant medications that prolong the QT/QTc interval.
11. Prior corticosteroid therapy within 14 days of first receipt of study drug.
12. Treatment with any investigational agent within 28 days of first receipt of study drug.
13. Acute or chronic infection. Any other diseases, metabolic dysfunction, physical examination finding, or clinical laboratory finding or any other medical condition that, in the opinion of the investigator, contraindicates the use of an investigational drug, or will impose excessive risk to the patient.
14. Known Human Immunodeficiency Virus (HIV), Hepatitis B Virus (HBV), or Hepatitis C Virus (HCV) infection.
15. History of clinically significant bowel disease including abdominal fistula, gastro-intestinal perforation, and diverticulitis.
16. Major surgery within 28 days of first receipt of study drug.
17. Pregnant or lactating women
18. Altered mental status or psychiatric disorder that, in the opinion of the investigator, would preclude a valid patient informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2010-08; Primary Completion 2012-11 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Occurrence of dose limiting toxicities | Upon completion of the study
Preliminary anti-tumour activity | Upon completion of the study

SECONDARY OUTCOMES:
To determine the pharmacokinetics of CH5132799 | Upon completion of the study
To characterise the pharmacodynamic effect of CH5132799 in surrogate tissues | Upon completion of the study

CONTACTS AND LOCATIONS:
Locations (1):
- Investigator Sites, London, Leeds, United Kingdom